CLINICAL TRIAL: NCT06816251
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of HRS-1893 in Non-Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Phase II Clinical Study of HRS-1893 in Non-obstructive Hypertrophic Cardiomyopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-1893-202
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Non-obstructive Hypertrophic Cardiomyopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-1893 low-dose group (Experimental)
  Interventions: Drug: HRS-1893
- HRS-1893 placebo low-dose group (Placebo Comparator)
  Interventions: Drug: HRS-1893 placebo
- HRS-1893 high-dose group (Experimental)
  Interventions: Drug: HRS-1893
- HRS-1893 placebo high-dose group (Placebo Comparator)
  Interventions: Drug: HRS-1893 placebo

INTERVENTIONS:
Drug: HRS-1893 — HRS-1893 tablet.
  Arms: HRS-1893 high-dose group; HRS-1893 low-dose group
Drug: HRS-1893 placebo — HRS-1893 tablet placebo.
  Arms: HRS-1893 placebo high-dose group; HRS-1893 placebo low-dose group

SUMMARY:
This study mainly evaluated the safety and tolerability of HRS-1893 in subjects with non-obstructive hypertrophic cardiomyopathy, and the efficacy and plasma concentrations of different dosing regimens in subjects with non-obstructive hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~85 years old (including boundary value), male or female.
2. Body mass index < 35 kg/m2.
3. Understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent form in writing.
4. Female subjects of childbearing potential must have a serum pregnancy test prior to the first dose with a negative result and must be non-lactating during the study.
5. Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to refrain from donating sperm/eggs from the time of signing the informed consent form until 3 months after the last dose of the trial drug, and comply with the relevant contraceptive requirements.

Exclusion Criteria:

1. Known or suspected infiltration, hereditary, or storage disorder that can cause myocardial hypertrophy.
2. Paroxysmal atrial flutter or atrial fibrillation with clinical symptoms at screening.
3. History of syncope or sustained ventricular tachycardia within 6 months prior to screening.
4. Those who have participated in the clinical trial of any drug or medical device within 3 months before screening.
5. Other conditions that the investigator considers the subject to be unsuitable for participating in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 14 weeks.
The incidence of left ventricular ejection fraction (LVEF) < 50% | Up to 14 weeks.

SECONDARY OUTCOMES:
Peak oxygen uptake (pVO2) value | About 12 weeks.
The cardiac troponin value | About 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided